Original Title: Owning Rights and Protection: GBV Prevention, Mitigation, and Response in Colombia (2023-2025)

Date of Document: February 27, 2024

NCT Number: Not currently available

### **ATTACHMENTS**

## <u>Informed consent document - English</u>

# ADULT CONSENT FORM — Owning Rights and Protection: GBV Prevention, Mitigation, and Response in Colombia (2023-2025) (ADULTS 18+ YEARS)

#### **Informed Consent Form**

the Passarcher socking consent: This form is to be used in asking for the consent of

| women 18 years and older to participate in the study. |
|---|
| Greeting |
| Hello, my name is May I please speak to you? |
| As I said, my name is We have come to speak with you because we would like to learn more about how to improve our entrepreneurship training program for women. We would like to learn more about your experiences before and after participating in the entrepreneurship training to make sure that we design and deliver the program in a way that will be successful. You are being invited to participate in this research because you meet the criteria outlined for participating in the HIAS program. |
| Background of research |
| Now I am going to describe the research activities, and your rights and responsibilities if you decide to take part. Please ask any questions about this research, including anything else about the research or this form that is not clear to you. Most importantly, know that you are allowed to say "no" to answering any questions, or stop participating at any time, and you will still be able to access HIAS services you are receiving now or in the future. |

We have come to speak with you because HIAS is conducting a study to better understand how its programs might help women in your community. If you choose to participate in this study, we will ask you some questions now as well as potentially two more times in the next year. You may also be assigned to participate in a livelihoods intervention according to the research procedure which involves randomization. However, non-selection for the research does not prevent you from later participation in HIAS programs. You are welcome to take part in other HIAS activities and if you are not selected for this livelihoods intervention, you may be provided with a referral for other programs.

# **Purpose of research**

We have come to speak with you because HIAS is working on improving its programming for women in this community and wants to know more about how this program might affect women's wellbeing, livelihood, and self-reliance. The reason we are here is to learn about a range of issues that women, like you, may experience. For example, we would like to ask some questions about your interpersonal skills such as communication, leadership, problem solving. We will also ask some questions about your perceptions related to economic wellbeing, employment and self-reliance. We know that you may experience a

number of different challenges living here, and we will ask you some questions about those experiences and challenges.

As I mentioned, you will be asked questions today by a study team member using a tablet. We may also visit you twice more in the next year to ask additional questions.

#### **Voluntary Participation**

There is no pressure on you to talk with us. You are free to say "No" and we will not be offended if you say you do not want to talk with us. Also, if you agree to talk with us, you are free at any time to decide not to answer any particular questions or to end the interview.

So I would like to ask permission to ask you survey questions for around 60-90 minutes. At any point of the discussion or activity, if you do not want to continue, you can tell us and we will stop. That is fine. You can also decide not to answer any questions at any time. None of these decisions will change the services you or your family receive here.

The survey data will be stored in a safe place with no mention of your name, and it will be destroyed once the study is completed.

#### **Benefits and Risks**

You will not receive any benefits, like money or other material benefits, by taking part in this research. However, as I mentioned, you may be randomly assigned to participate in a livelihoods intervention. What you tell us will help us understand how to improve this training for women like you in the future.

For this study, there is a risk that you may feel embarrassed or uncomfortable during the activity or discussion. Remember, if you are uncomfortable with any question or topic simply tell us that you do not want to discuss it and we will move on. If you are feeling sad or upset after the activity or discussion, you can tell us and we will find someone for you to talk to.

### Confidentiality

The information you give will be used only by Los Andes University, Washington University in St. Louis, and HIAS, and only for the purpose of research. All of the information that you provide will be kept confidential.

We will not share any information or answers with any of your family members or community members. Only our research staff will have access to your answers, and your identity will not be disclosed when data is shared with other researchers or when this study is published. For record-keeping purposes only, we have assigned you a unique study identification number. Only this number appears on our research documents; we will not put your name on these documents. Also, the interviews will be kept on a password-protected computer to which only the research staff will have access.

## **Additional Information**

If you have questions about the research, please contact Marcela Venegas by email at <a href="marcela.venegas@hias.org">marcela.venegas@hias.org</a>, or Arturo Harker, Universidad de los Andes focal point, at <a href="marcela.venegas@hias.org">a.harker@uniandes.edu.co</a> or +57-3107551902.

If you have questions about your rights as a subject in this research, please contact the IRB COMMITTEE: Research Ethics Committee of the Universidad de los Andes: <a href="mailto:comite-etica-investigaciones@uniandes.edu.co">comite-etica-investigaciones@uniandes.edu.co</a>.

Please feel free to take note of this information for future reference.

## **Informed Consent**

I will now ask you to show that you have heard about this research, from me, including the reason for the research, the activities, and the risks, benefits and alternatives. Please tell me now if you are willing to participate in this study. (If 'Yes,' apply thumbprint or signature.)

| Thank you for listening to me. |
|---|
| PARTICIPANT'S NAME (Print Name): |
| [ ] DOES NOT AGREE TO PARTICIPATE. (THANK PARTICIPANT FOR HIS/HER TIME AND END.) |
| [ ] AGREES TO PARTICIPATE. |
| [ ] AGREES TO AUDIO-RECORDING. |
| Name of Researcher Obtaining Consent: |
| Signature: |
| Date: |